CLINICAL TRIAL: NCT05624151
Title: Dexmedetomidine Versus Magnesium Sulphate Added to Bupivacaine in Infraorbital Nerve Block for Perioperative Analgesia in Paediatric Patients for Cleft Lip Surgery: A Prospective, Randomized Double Blinded Study
Brief Title: Dexmedetomidine Versus Magnesium Sulphate Added to Bupivacaine in Infraorbital Nerve Block for Perioperative Analgesia in Paediatric Patients for Cleft Lip Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R176/2022
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Magnesium Sulfate; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- general anesthesia+ infraorbital nerve block by dexmedetomidine plus bupivacaine (Active Comparator)
  Interventions: Drug: Dexmedetomidine +Bupivacaine
- general anesthesia+ infraorbital nerve block by magnesium sulphate plus bupivacaine (Active Comparator)
  Interventions: Drug: Magnesium Sulfate + Bupivacaine
- general anesthesia+infraorbital nerve block by bupivacaine only (Active Comparator)
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine +Bupivacaine — infraorbital nerve block by dexmedetomidine plus bupivacaine
  Arms: general anesthesia+ infraorbital nerve block by dexmedetomidine plus bupivacaine
Drug: Magnesium Sulfate + Bupivacaine — infraorbital nerve block by magnesium sulphate plus bupivacaine
  Arms: general anesthesia+ infraorbital nerve block by magnesium sulphate plus bupivacaine
Drug: Bupivacaine — infraorbital nerve block by bupivacaine only
  Arms: general anesthesia+infraorbital nerve block by bupivacaine only

SUMMARY:
Regional analgesia is considered the cornerstone for postoperative analgesia in paediatric patients. One of the most common birth defects which require surgical intervention early in life is the cleft lip. Infraorbital nerve block (IONB) has been used for postoperative analgesia in this delicate and sensitive area.

As the assessment of pain may be very challenging especially in young children, the local anaesthetics administration can be a safe alternative to opioids.[2] However, the regional block after a single dose of local anaesthetic is of limited duration and efficacy. Hence, the coadministration of adjuvants with local anaesthetics may be helpful for potentiation of analgesic effect.

Infraorbital nerve block is a well-recognized regional anaesthetic technique which can provide intraoperative and postoperative pain relief in nasal endoscopic surgery and in some types of oral and dental surgery including cleft lip repair . The block may also be used to help diagnose neuralgia arising from the second division of the trigeminal nerve. The technique for infraorbital nerve blockade is most performed as it exits the infraorbital foramen just below the inferior orbital rim.Dexmedetomidine (DE) is a potent α2 adrenoreceptor agonist and it is highly selective for α2 adrenoreceptor seven times more than clonidine. Many studies documented a prolonged duration and rapid onset of sensory block with the perineural injection of DE. Dexmedetomidine has been introduced as an adjuvant to local anaesthetics in both neuroaxial and peripheral nerve blocks. [9, 10] perineural dexmedetomidine has shown to prolong the duration of postoperative analgesia in addition to reducing the opioid consumption. The exact mechanism of peripheral nerve block produced by α2 adrenoreceptor agonists includes central analgesia, anti-inﬂammatory effect.Another suggested mechanism is that DE may exert its action through blocking the hyperpolarization-activated cation current after the transient sodium influx. The effect of magnesium was first recognized for the treatment of arrhythmia and preeclampsia, and its effect on anaesthesia and analgesia has recently been recognized. Magnesium sulphate has also been used as an adjunct to anaesthesia in recent years. It is also an effective analgesic agent for perioperative pain. Research have also reported that the intraoperative use of magnesium is characterized by a reduced use of anaesthetics and muscle relaxants. Furthermore, opioid use, postoperative nausea and vomiting, hypertension, and shivering have met a decreased trend with the use of magnesium sulphate. In a study performed by (El-Emam and El motlb) in 2019 they compared the efficacy of dexamethasone versus dexmedetomidine as an adjuvant to bupivacaine in ultrasound guided infraorbital nerve block in paediatric patients scheduled for cleft lip repair. they noticed that dexmedetomidine produced a more prolonged duration of analgesia and a lower pain score and increased sedation than produced by dexamethasone. Also, they found that Both dexamethasone and dexmedetomidine were tolerable with no significant difference regarding the incidence of postoperative nausea and vomiting or intraoperative hemodynamic changes.Aim of the work:

The purpose of this randomized controlled double-blind study is to compare the efficacy of Dexmedetomidine or Magnesium sulphate as adjuvants for bupivacaine in infraorbital nerve block in paediatric patients scheduled for cleft lip repair.

ELIGIBILITY:
Inclusion Criteria:

* patients who will be scheduled for indicated cleft lip surgery. • physical status American Society of Anesthesiologists (ASA) I or II.

Exclusion Criteria:

* failure to gain the consent from parents
* allergy to any of drugs used
* coagulopathy
* thrombocytopenia
* history of any lower or upper airway disorders
* history of sleep apnea syndrome with a suspected need for postoperative ventilation
* any wound or infection related to puncture site
* major illness failure to gain the consent of parents.

Ages: 3 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
first time to analgesic requirment | 1st 24 hour
  paracetamol will be given as the first rescue analgesia

SECONDARY OUTCOMES:
Total amount of analgesics | 1st 24 hours postoperatively
pain score (FLACC Score) face, leg , cry, activity ,conslolability | 1st 24 postoperatively
  assess pain in patients (ranging from 0-10, where 0 = no pain, 10 = worst pain)
postoperative side effects | 1st 24 hour postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt